CLINICAL TRIAL: NCT01755052
Title: SILVER-AMI: Risk Stratification in Older Persons With Acute Myocardial Infarction
Brief Title: SILVER-AMI: Outcomes in Older Persons With Heart Attacks
Acronym: SILVER-AMI
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1205010311; 1R01HL115295-01 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-12-21 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Geriatrics; Cardiology; Aging; Heart Attack; Risk Factors; Quality of Care; Risk Models
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SILVER-AMI is a research study of older persons who are admitted to the hospital with a heart attack. Patients will be interviewed in the hospital and again 6 months later. The researchers will also collect detailed medical record information to understand the effect of heart attacks on older persons.

The research team at Yale University will use this information to develop a risk model that can be used to help doctors predict recovery. The goal of the study is to help older people in the future make well-informed decisions about their health care during a heart attack.

DETAILED DESCRIPTION:
The overall objective of this study is to develop and validate risk stratification tools for older adults who have recently had an Acute Myocardial Infarction (AMI). While there is emerging interest in understanding the role of geriatric conditions as they pertain to cardiovascular outcomes, there is no standard, feasible assessment of older patients with AMI that can stratify their risk of subsequent morbidity and mortality. Currently available risk models are designed solely to predict clinical events (e.g. mortality, reinfarction). This is insufficient for shared decision making with older patients, who consistently rate maintenance of favorable health status as a top priority. This study will address these gaps by melding principles from geriatrics and cardiology to create post-AMI risk models specifically designed for older patients. This study is significant because older persons with AMI are a growing, yet understudied, population.

Dr. Sarwat Chaudhry at Yale University is conducting a multi-center, observational study designed to collect data about the post-AMI recovery period that will be used to generate risk models for older patients with AMI. The intent of the study is to use the knowledge from the data collected in SILVER-AMI to ultimately design interventions to improve the care and outcomes of older patients with AMI.

Study coordinators will screen older patients hospitalized with an AMI. Participants will be assessed at baseline prior to AMI hospital discharge through an interview, physical assessment and medical record review. One follow-up interview will be conducted approximately 6 months later by the Yale Follow-up Center. Clinical outcomes will be assessed for the follow-up period occurring 6 months post AMI hospitalization through self-report and medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥75 years upon admission to the hospital
2. Elevation of cardiac markers within 24 hours of presentation to the hospital

   a. Troponin must rise above the upper limit of normal established by the hospital as a determinate of cardiac injury.
3. Any one of the following:

   1. Symptoms of ischemia
   2. ECG with ischemic changes
   3. Imaging evidence of Infarction
   4. Intracoronary thrombus on angiography

Exclusion Criteria:

1. Patient transferred from another hospital with a length of stay >48 hours at the referring hospital.
2. Refused Informed Consent
3. Decisional impairment with no legally authorized representative
4. AMI is secondary to chest trauma
5. AMI is secondary to in-patient procedure or surgery
6. History of heart transplant
7. Non-English/Non-Spanish speaking
8. Inability to complete interview (e.g. comatose or aphasia)
9. Inability to contact for follow-up (e.g. no access to phone, not living in the country)
10. Currently a prisoner
11. Death prior to enrollment
12. Previously enrolled in SILVER-AMI
13. Troponin elevation is the result of apical ballooning syndrome (i.e., Takotsubo)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults admitted to the hospital with a heart attack
Sampling Method: Non-Probability Sample
Enrollment: 3042 (Actual)
Dates: Start 2013-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
All-cause hospital readmission | up to six months

SECONDARY OUTCOMES:
All-cause mortality | Up to six months
Decline in health status | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Sarwat Chaudhry, MD, Principal Investigator — Yale University
Locations (81):
- United States (81):
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Los Alamitos Internal Medical Group, Los Alamitos, California
  - Mercy General Hospital, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - St. Joseph's Medical Center, Stockton, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - The Danbury Hospital and the Western Connecticut Medical, Danbury, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Florida Hospital Pepin Heart Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - The Corporation of Mercer University, Macon, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University Of Chicago, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - St. Francis Medical Group, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Meritus Medical Center, Hagerstown, Maryland
  - Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - McLaren Cardiovascular Group, Okemos, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mid America Heart Institute St. Luke's Hospital, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - The International Heart Institute of Montana, Missoula, Montana
  - Nebraska Specialty Network, Lincoln, Nebraska
  - CHI-Health-Alegent Creighton Research, Omaha, Nebraska
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - New York University School of Medicine, New York, New York
  - The Trustees of Columbia University in the City of New York, New York, New York
  - St. Francis Research & Educational Corporation, Roslyn, New York
  - The Research Foundation for the State University of New York, Stony Brook, New York
  - Montefiore/Albert Einstein Medical Center, The Bronx, New York
  - Mission Medical Associates, Inc. dba Asheville Cardiology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Research, Fargo, North Dakota
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Good Samaritan Hospital, Corvallis, Corvallis, Oregon
  - Providence Health & Services, Portland, Oregon
  - OHSU: Oregon Health & Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Inc., Rapid City, South Dakota
  - Providence Healthcare Network, Waco, Texas
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Sentara Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - St Mary's Medical Center, Huntington, West Virginia
  - Bellin Memorial Hospital, Inc., Green Bay, Wisconsin
  - Aurora Research Institute, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Dodson JA, Hajduk AM, Geda M, Krumholz HM, Murphy TE, Tsang S, Tinetti ME, Nanna MG, McNamara R, Gill TM, Chaudhry SI. Predicting 6-Month Mortality for Older Adults Hospitalized With Acute Myocardial Infarction: A Cohort Study. Ann Intern Med. 2020 Jan 7;172(1):12-21. doi: 10.7326/M19-0974. Epub 2019 Dec 10. PMID 31816630
- [Derived] Dodson JA, Hajduk AM, Murphy TE, Geda M, Krumholz HM, Tsang S, Nanna MG, Tinetti ME, Goldstein D, Forman DE, Alexander KP, Gill TM, Chaudhry SI. Thirty-Day Readmission Risk Model for Older Adults Hospitalized With Acute Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005320. doi: 10.1161/CIRCOUTCOMES.118.005320. PMID 31010300
- [Derived] Dodson JA, Geda M, Krumholz HM, Lorenze N, Murphy TE, Allore HG, Charpentier P, Tsang SW, Acampora D, Tinetti ME, Gill TM, Chaudhry SI. Design and rationale of the comprehensive evaluation of risk factors in older patients with AMI (SILVER-AMI) study. BMC Health Serv Res. 2014 Nov 5;14:506. doi: 10.1186/s12913-014-0506-4. PMID 25370536